CLINICAL TRIAL: NCT02691611
Title: Defining Epigenetic Regulation of Immunity in Alpha-1 Anti-trypsin Deficiency
Brief Title: Epigenetic Regulation of Immunity in Alpha-1 Anti-trypsin Deficiency
Acronym: AATD_Epi
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: HS-2939
Record Dates: First submitted 2016-02-12; First posted 2016-02-25 (Estimated); Last update posted 2025-06-06 (Actual); Status verified 2019-03

CONDITIONS: Alpha 1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Alpha-1 Antitrypsin: All AATD patients who will start treatment with alpha-1 antitrypsin augmentation therapy
- Healthy Control: Healthy controls with no lung diseases

SUMMARY:
The investigators hypothesize that environmentally influenced histone modifications regulate AM mediated inflammation, contributing to a variable clinical course of AATD, and may also influence or be influenced by the activity of AAT augmentation therapy.

DETAILED DESCRIPTION:
The variable natural clinical course of alpha-1 anti-trypsin deficiency (AATD) disease and strong influence of environmental exposures such as smoking, implicate a major role for epigenetic mechanisms in modifying AATD disease penetrance. The goal of this study proposal is to investigate epigenetic regulation of alveolar macrophage (AM) inflammation and function in AATD homozygous alpha 1-protease inhibitor deficiency (PiZZ) (two Z genes) and homozygous alpha 1-protease inhibitor deficiency (PiMZ) (one M and one Z gene) patients. The investigators proposal focuses on epigenetic histone modifications and gene expression specifically in AM.

AAT augmentation therapy, which alters disease symptoms, may also modulate AM epigenetics. To identify epigenetic regulation of AM inflammation in AATD in the context of AAT therapy, the investigators will perform and computationally integrate chromatin immunoprecipitation sequencing (ChIP-seq) and RNA-seq data. This will help elucidate the immunomodulatory mechanisms regulating AATD and provide an epigenetic map for diagnosis and targeted treatment. The investigators will test the efficacy of FDA-approved histone modifying drugs, such as Suberoylanilide Hydroxamic Acid (SAHA) and more specific next-generation histone modifiers, such as GSK-J4, to modulate AM AATD-associated activity ex vivo.

The goal of this study is to enroll up to a total of 13 AATD cases and 6 healthy controls. All AATD patients will be asked to give a blood sample and/or undergo a bronchoscopy. AATD patients will also be asked to undergo a follow up bronchoscopy and/or blood draw after 6 months if treatment with alpha-1 antitrypsin augmentation therapy is initiated to study the changes in these markers after augmentation therapy.

ELIGIBILITY:
Inclusion Criteria:

AATD

* Age between the ages of 18 and 85
* Have a diagnosis of AATD PiZZ or PiMZ established by AAT blood levels and Pi genotyping
* Are not and have not been on AAT augmentation therapy for the past 6 months
* Able to tolerate and willing to undergo study procedures
* Provide signed informed consent.

Exclusion Criteria:

AATD

1. History of comorbid condition severe enough to significantly increase risks based on investigator discretion
2. Diagnosis of unstable cardiovascular disease including myocardial infarction in the past 6 weeks, uncontrolled congestive heart failure, or uncontrolled arrhythmia
3. Partial Pressure of Oxygen (PaO2) on room air at rest <50 mmHg or Oxygen saturation (SaO2) on room air at rest <85%
4. Post bronchodilator Forced expiratory volume in one second (FEV1)<30% predicted
5. Use of anticoagulation (patients on warfarin or clopidogrel will be excluded; patients on aspirin alone can be studied even with concurrent use)
6. Dementia or other cognitive dysfunction which in the opinion of the investigator would prevent the participant from consenting to the study or completing study procedures
7. Active pulmonary infection with tuberculosis
8. History of pulmonary embolism in the past 2 years
9. Non-Chronic Obstructive Pulmonary Disease (COPD) obstructive disease (various bronchiolitides, sarcoid, lymphangioleiomyomatosis (LAM), histiocytosis X) or parenchymal lung disease, pulmonary vascular disease, pleural disease, severe kyphoscoliosis, neuromuscular weakness, or other cardiovascular and pulmonary disease, that, in the opinion of the investigator, limit the interpretability of the pulmonary function measures
10. Prior significant difficulties with pulmonary function testing
11. Hypersensitivity to or intolerance of albuterol sulfate or ipratropium bromide or propellants or excipients of the inhalers
12. Hypersensitivity to or intolerance of all drugs required for sedation during conscious sedation bronchoscopy.
13. History of Lung volume reduction surgery, lung resection or bronchoscopic lung volume reduction in any form
14. History of lung or other organ transplant
15. History of large thoracic metal implants (e.g., Implantable cardioverter-defibrillator (AICD) and/or pacemaker) that in the opinion of the investigator limit the interpretability of CT scans
16. Currently taking >=10mg a day/20mg every other day of prednisone or equivalent systemic corticosteroid
17. Currently taking any immunosuppressive agent excepting systemic corticosteroids
18. History of lung cancer or any cancer that spread to multiple locations in the body
19. Current illicit substance abuse, excluding marijuana
20. Known HIV/AIDS infection
21. History of or current exposure to chemotherapy or radiation treatments that, in the opinion of the investigator, limits the interpretability of the pulmonary function measures.
22. Has a BMI > 40 kg/m2 at baseline exam
23. Current or planned pregnancy within the study course.
24. Currently institutionalized (e.g., prisons, long-term care facilities)
25. Have a genotype of PiMZ and ever received intravenous or inhaled alpha-1 augmentation therapy (Alpha-1 Proteinase Inhibitor, A1PI)

Conditional Exclusions

1. Participants who present with an upper respiratory infection or pulmonary exacerbation, either solely participant-identified or that has been clinically treated, in the last six weeks can be rescreened for the study once the six-week window has passed.
2. Participants who present with current use of acute antibiotics or steroids can be rescreened for the study ≥30 days after discontinuing acute antibiotics/steroids.

   This does not apply to participants who are on chronic prednisone therapy of <10 mg per day or <20 mg every other day.
3. Participants who present with a myocardial infarction or eye, chest, or abdominal surgery within six weeks can be rescreened after the six week window has passed.

   Study coordinators should consult with the site principal investigator prior to rescreening these participants.
4. Female participants who present <3 months after giving birth will be asked to reschedule their visit until three months have passed since the birth.
5. Individuals who are PiZZ receiving alpha-1 augmentation therapy (Alpha-1 Proteinase Inhibitor, A1PI) must be off augmentation therapy for >6 months to qualify for stratified enrollment in the PiZZ group not receiving augmentation therapy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * AATD from clinic
  * Healthy controls from community
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2015-12; Primary Completion 2018-11 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Epigenetic signature of specific inflammation-associated histone modifications from CD14+ macrophages | Change from Baseline histones at 6 months

SECONDARY OUTCOMES:
Epigenetically regulated genomic profile of AATD in AM | Change from Baseline polyA RNA at 6 months
Epigenetic mechanisms to regulate gene expression and cell function | Change from Baseline epigenetic modified cells at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Brian P O'Connor, PhD, Principal Investigator — National Jewish Health; Nabeel Y Hamzeh, MD, Principal Investigator — National Jewish Health; Robert Sandhaus, MD, PhD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silverman EK, Sandhaus RA. Clinical practice. Alpha1-antitrypsin deficiency. N Engl J Med. 2009 Jun 25;360(26):2749-57. doi: 10.1056/NEJMcp0900449. No abstract available. PMID 19553648
- [Background] Kim WJ, Wood AM, Barker AF, Brantly ML, Campbell EJ, Eden E, McElvaney G, Rennard SI, Sandhaus RA, Stocks JM, Stoller JK, Strange C, Turino G, Silverman EK, Stockley RA, Demeo DL. Association of IREB2 and CHRNA3 polymorphisms with airflow obstruction in severe alpha-1 antitrypsin deficiency. Respir Res. 2012 Feb 22;13(1):16. doi: 10.1186/1465-9921-13-16. PMID 22356581
- [Background] Bouchecareilh M, Hutt DM, Szajner P, Flotte TR, Balch WE. Histone deacetylase inhibitor (HDACi) suberoylanilide hydroxamic acid (SAHA)-mediated correction of alpha1-antitrypsin deficiency. J Biol Chem. 2012 Nov 2;287(45):38265-78. doi: 10.1074/jbc.M112.404707. Epub 2012 Sep 20. PMID 22995909
- [Background] Breton CV, Byun HM, Wenten M, Pan F, Yang A, Gilliland FD. Prenatal tobacco smoke exposure affects global and gene-specific DNA methylation. Am J Respir Crit Care Med. 2009 Sep 1;180(5):462-7. doi: 10.1164/rccm.200901-0135OC. Epub 2009 Jun 4. PMID 19498054
- [Background] Sanders YY, Ambalavanan N, Halloran B, Zhang X, Liu H, Crossman DK, Bray M, Zhang K, Thannickal VJ, Hagood JS. Altered DNA methylation profile in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2012 Sep 15;186(6):525-35. doi: 10.1164/rccm.201201-0077OC. Epub 2012 Jun 14. PMID 22700861
- [Background] Jeffries MA, Dozmorov M, Tang Y, Merrill JT, Wren JD, Sawalha AH. Genome-wide DNA methylation patterns in CD4+ T cells from patients with systemic lupus erythematosus. Epigenetics. 2011 May;6(5):593-601. doi: 10.4161/epi.6.5.15374. Epub 2011 May 1. PMID 21436623
- [Background] Cortessis VK, Thomas DC, Levine AJ, Breton CV, Mack TM, Siegmund KD, Haile RW, Laird PW. Environmental epigenetics: prospects for studying epigenetic mediation of exposure-response relationships. Hum Genet. 2012 Oct;131(10):1565-89. doi: 10.1007/s00439-012-1189-8. Epub 2012 Jun 28. PMID 22740325
- [Background] Akimova T, Beier UH, Liu Y, Wang L, Hancock WW. Histone/protein deacetylases and T-cell immune responses. Blood. 2012 Mar 15;119(11):2443-51. doi: 10.1182/blood-2011-10-292003. Epub 2012 Jan 12. PMID 22246031
- [Background] Jirtle RL, Skinner MK. Environmental epigenomics and disease susceptibility. Nat Rev Genet. 2007 Apr;8(4):253-62. doi: 10.1038/nrg2045. PMID 17363974
- [Background] Feinberg AP. Epigenetics at the epicenter of modern medicine. JAMA. 2008 Mar 19;299(11):1345-50. doi: 10.1001/jama.299.11.1345. PMID 18349095
- [Background] Fraga MF, Ballestar E, Paz MF, Ropero S, Setien F, Ballestar ML, Heine-Suner D, Cigudosa JC, Urioste M, Benitez J, Boix-Chornet M, Sanchez-Aguilera A, Ling C, Carlsson E, Poulsen P, Vaag A, Stephan Z, Spector TD, Wu YZ, Plass C, Esteller M. Epigenetic differences arise during the lifetime of monozygotic twins. Proc Natl Acad Sci U S A. 2005 Jul 26;102(30):10604-9. doi: 10.1073/pnas.0500398102. Epub 2005 Jul 11. PMID 16009939
- [Background] Miller RL, Ho SM. Environmental epigenetics and asthma: current concepts and call for studies. Am J Respir Crit Care Med. 2008 Mar 15;177(6):567-73. doi: 10.1164/rccm.200710-1511PP. Epub 2008 Jan 10. PMID 18187692
- [Background] Yang IV, Schwartz DA. Epigenetic control of gene expression in the lung. Am J Respir Crit Care Med. 2011 May 15;183(10):1295-301. doi: 10.1164/rccm.201010-1579PP. PMID 21596832
- [Background] Hutt DM, Herman D, Rodrigues AP, Noel S, Pilewski JM, Matteson J, Hoch B, Kellner W, Kelly JW, Schmidt A, Thomas PJ, Matsumura Y, Skach WR, Gentzsch M, Riordan JR, Sorscher EJ, Okiyoneda T, Yates JR 3rd, Lukacs GL, Frizzell RA, Manning G, Gottesfeld JM, Balch WE. Reduced histone deacetylase 7 activity restores function to misfolded CFTR in cystic fibrosis. Nat Chem Biol. 2010 Jan;6(1):25-33. doi: 10.1038/nchembio.275. Epub 2009 Dec 6. PMID 19966789
- [Background] Mizuno S, Yasuo M, Bogaard HJ, Kraskauskas D, Natarajan R, Voelkel NF. Inhibition of histone deacetylase causes emphysema. Am J Physiol Lung Cell Mol Physiol. 2011 Mar;300(3):L402-13. doi: 10.1152/ajplung.00207.2010. Epub 2010 Dec 17. PMID 21224215
- [Background] Chen X, Barozzi I, Termanini A, Prosperini E, Recchiuti A, Dalli J, Mietton F, Matteoli G, Hiebert S, Natoli G. Requirement for the histone deacetylase Hdac3 for the inflammatory gene expression program in macrophages. Proc Natl Acad Sci U S A. 2012 Oct 16;109(42):E2865-74. doi: 10.1073/pnas.1121131109. Epub 2012 Jul 16. PMID 22802645
- [Background] Szyf M. Epigenetics, DNA methylation, and chromatin modifying drugs. Annu Rev Pharmacol Toxicol. 2009;49:243-63. doi: 10.1146/annurev-pharmtox-061008-103102. PMID 18851683
- [Background] Natoli G, Testa G, De Santa F. The future therapeutic potential of histone demethylases: A critical analysis. Curr Opin Drug Discov Devel. 2009 Sep;12(5):607-15. PMID 19736620
- [Background] De Santa F, Narang V, Yap ZH, Tusi BK, Burgold T, Austenaa L, Bucci G, Caganova M, Notarbartolo S, Casola S, Testa G, Sung WK, Wei CL, Natoli G. Jmjd3 contributes to the control of gene expression in LPS-activated macrophages. EMBO J. 2009 Nov 4;28(21):3341-52. doi: 10.1038/emboj.2009.271. Epub 2009 Sep 24. PMID 19779457
- [Background] De Santa F, Totaro MG, Prosperini E, Notarbartolo S, Testa G, Natoli G. The histone H3 lysine-27 demethylase Jmjd3 links inflammation to inhibition of polycomb-mediated gene silencing. Cell. 2007 Sep 21;130(6):1083-94. doi: 10.1016/j.cell.2007.08.019. Epub 2007 Sep 6. PMID 17825402
- [Background] Kruidenier L, Chung CW, Cheng Z, Liddle J, Che K, Joberty G, Bantscheff M, Bountra C, Bridges A, Diallo H, Eberhard D, Hutchinson S, Jones E, Katso R, Leveridge M, Mander PK, Mosley J, Ramirez-Molina C, Rowland P, Schofield CJ, Sheppard RJ, Smith JE, Swales C, Tanner R, Thomas P, Tumber A, Drewes G, Oppermann U, Patel DJ, Lee K, Wilson DM. A selective jumonji H3K27 demethylase inhibitor modulates the proinflammatory macrophage response. Nature. 2012 Aug 16;488(7411):404-8. doi: 10.1038/nature11262. PMID 22842901
- [Background] Natoli G, Ghisletti S, Barozzi I. The genomic landscapes of inflammation. Genes Dev. 2011 Jan 15;25(2):101-6. doi: 10.1101/gad.2018811. PMID 21245163
- [Background] Bouchecareilh M, Balch WE. Proteostasis, an emerging therapeutic paradigm for managing inflammatory airway stress disease. Curr Mol Med. 2012 Aug;12(7):815-26. doi: 10.2174/156652412801318782. PMID 22697348
- [Background] DeMeo DL, Silverman EK. Alpha1-antitrypsin deficiency. 2: genetic aspects of alpha(1)-antitrypsin deficiency: phenotypes and genetic modifiers of emphysema risk. Thorax. 2004 Mar;59(3):259-64. doi: 10.1136/thx.2003.006502. PMID 14985567
- [Background] Demeo DL, Sandhaus RA, Barker AF, Brantly ML, Eden E, McElvaney NG, Rennard S, Burchard E, Stocks JM, Stoller JK, Strange C, Turino GM, Campbell EJ, Silverman EK. Determinants of airflow obstruction in severe alpha-1-antitrypsin deficiency. Thorax. 2007 Sep;62(9):806-13. doi: 10.1136/thx.2006.075846. Epub 2007 Mar 27. PMID 17389752
- [Background] Seersholm N, Kok-Jensen A, Dirksen A. Survival of patients with severe alpha 1-antitrypsin deficiency with special reference to non-index cases. Thorax. 1994 Jul;49(7):695-8. doi: 10.1136/thx.49.7.695. PMID 8066566
- [Background] Wolff GL, Kodell RL, Moore SR, Cooney CA. Maternal epigenetics and methyl supplements affect agouti gene expression in Avy/a mice. FASEB J. 1998 Aug;12(11):949-57. PMID 9707167
- [Background] Seersholm N, Wencker M, Banik N, Viskum K, Dirksen A, Kok-Jensen A, Konietzko N. Does alpha1-antitrypsin augmentation therapy slow the annual decline in FEV1 in patients with severe hereditary alpha1-antitrypsin deficiency? Wissenschaftliche Arbeitsgemeinschaft zur Therapie von Lungenerkrankungen (WATL) alpha1-AT study group. Eur Respir J. 1997 Oct;10(10):2260-3. doi: 10.1183/09031936.97.10102260. PMID 9387950
- [Background] Wencker M, Fuhrmann B, Banik N, Konietzko N; Wissenschaftliche Arbeitsgemeinschaft zur Therapie von Lungenerkrankungen. Longitudinal follow-up of patients with alpha(1)-protease inhibitor deficiency before and during therapy with IV alpha(1)-protease inhibitor. Chest. 2001 Mar;119(3):737-44. doi: 10.1378/chest.119.3.737. PMID 11243951
- [Background] Stockley RA, Bayley DL, Unsal I, Dowson LJ. The effect of augmentation therapy on bronchial inflammation in alpha1-antitrypsin deficiency. Am J Respir Crit Care Med. 2002 Jun 1;165(11):1494-8. doi: 10.1164/rccm.2109013. PMID 12045122
- [Background] Dirksen A, Piitulainen E, Parr DG, Deng C, Wencker M, Shaker SB, Stockley RA. Exploring the role of CT densitometry: a randomised study of augmentation therapy in alpha1-antitrypsin deficiency. Eur Respir J. 2009 Jun;33(6):1345-53. doi: 10.1183/09031936.00159408. Epub 2009 Feb 5. PMID 19196813
- [Background] Gottlieb DJ, Luisetti M, Stone PJ, Allegra L, Cantey-Kiser JM, Grassi C, Snider GL. Short-term supplementation therapy does not affect elastin degradation in severe alpha(1)-antitrypsin deficiency. The American-Italian AATD Study Group. Am J Respir Crit Care Med. 2000 Dec;162(6):2069-72. doi: 10.1164/ajrccm.162.6.2002032. PMID 11112116
- [Background] Teckman JH, Jain A. Advances in alpha-1-antitrypsin deficiency liver disease. Curr Gastroenterol Rep. 2014 Jan;16(1):367. doi: 10.1007/s11894-013-0367-8. PMID 24338605